CLINICAL TRIAL: NCT01750697
Title: A Phase IIA, International, Multicenter, Open-label, Uncontrolled Study to Evaluate The Safety And Pharmacokinetics of 4 × 375 mg/m2 Intravenous Rituximab in Pediatric Patients With Severe Granulomatosis With Polyangiitis (Wegener's) or Microscopic Polyangiitis
Brief Title: A Phase IIa Study of Intravenous Rituximab in Pediatric Participants With Severe Granulomatosis With Polyangiitis (Wegener's) or Microscopic Polyangiitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WA25615; 2012-002062-13 (EudraCT Number)
Record Dates: First submitted 2012-12-13; First posted 2012-12-17 (Estimated); Results first posted 2019-06-26 (Actual); Last update posted 2019-06-26 (Actual); Status verified 2019-06

CONDITIONS: Granulomatosis With Polyangiitis
MeSH Terms: conditions — Granulomatosis with Polyangiitis | interventions — Rituximab

ARMS (1):
- Rituximab (Experimental)
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Participants will receive rituximab 375 mg/m^2 IV infusion on Days 1, 8, 15 and 22. Rituximab infusions will be given at a rate of 25 milligrams per hour (mg/h). This may be escalated at a rate of 25 mg/h increments every 30 minutes to a maximum of 200 mg/h.
  Other Names: MabThera/Rituxan

SUMMARY:
This Phase IIa international multicenter, open-label, uncontrolled study will evaluate the safety and pharmacokinetics of rituximab (MabThera/Rituxan) in pediatric participants with severe granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA). Participants will receive rituximab 375 milligrams per square meter (mg/m^2) intravenously (IV) on Days 1, 8, 15 and 22.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of GPA (EULAR/PRINTO/PRES 2008, Ankara criteria for childhood Wegener's granulomatosis) or diagnosis of MPA (according to the Chapel Hill Consensus Conference)
* Newly diagnosed participants or participants with relapsing disease according to the following definition:

The recurrence or new onset of potentially organ- or life-threatening disease (i.e. one or more major Birmingham Vasculitis Activity Score for Wegener's Granulomatosis [BVAS/WG] items or disease severe enough to require treatment with cyclophosphamide)

* For participants of reproductive potential (males and females), use of reliable means of contraception throughout the study participation
* For all eligible participants mandatory prophylactic treatment for Pneumocystis jirovecii infection

Exclusion Criteria:

* Diagnosis of Churg-Strauss syndrome, as defined by the Chapel Hill Consensus Conference
* Limited disease that would not normally be treated with cyclophosphamide
* Severe disease requiring mechanical ventilation due to alveolar hemorrhage
* Requirement for plasmapheresis or dialysis at screening
* Incomplete recovery from recent surgery or less than (<) 12 weeks since surgery prior to baseline or planned within 24 weeks of baseline
* Lack of peripheral venous access
* Pregnancy or breast-feeding
* Evidence of other significant uncontrolled concomitant disease, or of disorder or condition that, in the investigator's opinion, would preclude or interfere with participation of participant
* Primary or secondary immunodeficiency (history of or currently active), including known history of human immunodeficiency virus (HIV) infection
* Evidence of active tuberculosis (participants receiving chemoprophylaxis for latent tuberculosis infection are eligible for the study)
* Known active infection of any kind (excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization or treatment with IV anti-infective agents within 4 weeks of baseline or completion of oral anti-infective agents within 2 weeks prior to baseline. Entry into this study may be reconsidered once the infection has fully resolved
* History of deep space/tissue infection within 24 weeks prior to baseline
* History of serious recurrent or chronic infection
* History of cancer (except for basal cell and squamous cell carcinoma of the skin that have been excised and cured)
* Currently active alcohol or drug abuse or history of alcohol or drug abuse
* History of severe allergic or anaphylactic reaction to a biologic agent or known hypersensitivity to any component of rituximab or to murine proteins
* Treatment with rituximab or other biologic B cell-targeted therapy (e.g., anti- Cluster of Differentiation [CD] 19, anti-CD20, anti-CD22, or anti-B-lymphocyte stimulator [BLys]/B-cell activating factor [BAFF]) within 6 months prior to baseline visit
* Previous treatment with an anti-alpha 4 integrin antibody or co-stimulation modulator
* Previous treatment with other cell-depleting therapies, including, but not limited to, investigational agents (e.g., alemtuzumab, anti-CD4, anti-CD5, anti-CD3, and anti-CD11a)
* Receipt of oral or IV cyclophosphamide within the previous 4 months prior to the baseline visit
* Receipt of infliximab within 3 months, adalimumab within 2 months or etanercept within 1 month prior to the baseline visit
* Treatment with any investigational agent within 28 days of baseline or 5 half-lives of the investigational drug (whichever is longer)
* Receipt of any live attenuated vaccine within 28 days prior to baseline
* Intolerance or contraindications to IV glucocorticoids
* Positive serum human chorionic gonadotropin measured at screening or a positive pregnancy test prior to the first rituximab infusion for participants of childbearing potential
* Positive tests for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (HBcAb), hepatitis B virus (HBV), or hepatitis C serology
* Level of Immunoglobulin (Ig) M below lower limit of normal of age-specific reference range
* Level of IgG below 5.65 milligram per milliliter
* Absolute neutrophil count < 1.5 × 10^3 per microliter and platelet count < 130 × 10^3 per microliter
* Estimated Glomerular Filtration Rate < 15 milliliter per minute per 1.73 m^2
* Alanine aminotransferase or aspartate aminotransferase levels greater than 2.5 times the upper limit of normal (for age and sex) that cannot be attributed to underlying granulomatosis with polyangiitis (GPA) or microscopic polyangiitis (MPA)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2013-05-23 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2018-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (23):
- United States (6):
  - University of Louisville Research Foundation, Inc; Kosair Charities Pediatric Clinical Research Unit, Louisville, Kentucky
  - Hackensack University Medical Center, Hackensack, New Jersey
  - COLUMBIA PRESBYTERIAN MEDICAL CENTER, Research Pharmacy, William Black Medical Research Building, New York, New York
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - The Cleveland Clinic Foundation; Rheumatic and Immunologic Diseases, Cleveland, Ohio
  - University of Utah; Immunology/Rheumatology/Allergy, Salt Lake City, Utah
- Canada (3):
  - Alberta Children'S Hospital, Calgary, Alberta
  - Children's and Women's Health Center / BC Children's Hospital, Vancouver, British Columbia
  - The Hospital for Sick Children Research Institute, Toronto, Ontario
- France (2):
  - Hopital Femme Mere Enfant; Ped Nephrologie Rhumatologie, Bron
  - Hop Necker Enfants Malades;UIH, Paris
- Germany (2):
  - Universitätsklinikum für Kinder und Jugendmedizin Hamburg, Hamburg
  - KfH-Nierenzentrum fur Kinder und Jugendliche, Heidelberg
- Italy (3):
  - Irccs Ospedale Pediatrico Bambin Gesu - Dip. Di Medicina, Rome, Lazio
  - Istituto Giannina Gaslini-Ospedale Pediatrico IRCCS, Genoa, Liguria
  - Univ. Di Padova - Dip. Di Pediatria - Unita' Reumatol. Pediatrica, Padua, Veneto
- Serbia (2):
  - Childrens University Hospital, Belgrade
  - Clinical Center Nis, Niš
- Turkey (Türkiye) (2):
  - Hacettepe University, School of Medicine; Pediatrics Department, Ankara
  - Istanbul University, Cerrahpasa Medical Faculty; Pediatrics Department, Istanbul
- United Kingdom (3):
  - Alder Hey Children s Hospital; Department of Pediatrics, Liverpool
  - Great Ormond Street Children's Hospital; Centre of Paediatric & Adolescent Rheumatology, London
  - Nottingham Children's Hospital, Nottingham

REFERENCES:
- [Derived] Melega S, Brogan P, Cleary G, Hersh AO, Kasapcopur O, Rangaraj S, Yeung RSM, Zeft A, Cooper J, Pordeli P, Kirchner P, Lehane PB. Evaluation of Serious Infection in Pediatric Patients with Low Immunoglobulin Levels Receiving Rituximab for Granulomatosis with Polyangiitis or Microscopic Polyangiitis. Rheumatol Ther. 2022 Apr;9(2):721-734. doi: 10.1007/s40744-022-00433-0. Epub 2022 Mar 12. PMID 35279811
- [Derived] Brogan P, Yeung RSM, Cleary G, Rangaraj S, Kasapcopur O, Hersh AO, Li S, Paripovic D, Schikler K, Zeft A, Bracaglia C, Eleftheriou D, Pordeli P, Melega S, Jamois C, Gaudreault J, Michalska M, Brunetta P, Cooper JC, Lehane PB; PePRS Study Group. Phase IIa Global Study Evaluating Rituximab for the Treatment of Pediatric Patients With Granulomatosis With Polyangiitis or Microscopic Polyangiitis. Arthritis Rheumatol. 2022 Jan;74(1):124-133. doi: 10.1002/art.41901. Epub 2021 Dec 5. PMID 34164952

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 25 participants were enrolled in the study over a 3.5 year period from 11 sites across the United Kingdom, Italy, Serbia, Turkey, Canada and the United States.
Pre-assignment Details: The screening visit occurred up to 28 days prior to the Day 1 baseline visit. Following successful screening, eligible participants entered the 6 month Remission Induction Phase of the study.
Groups:
- Rituximab: Participants received rituximab as an intravenous (IV) infusion of 375 milligrams per meter squared (mg/m^2) once a week on Days 1, 8, 15 and 22 during the Remission Induction Phase (Day 1 (baseline) to Month 6) and were followed for a minimum of 18 months (maximum 4.5yrs) during the Follow-up Phase until the Common-closeout (CCO))
Period: Overall Study
Arm/Group | Rituximab
Started (Remission Induction Phase (Day 1 to Month 6)) | 25
Completed (Remission Induction Phase (Day 1 to Month 6)) | 25
Follow-up Phase ((Month 6 to Month 18)) | 24 (Completed required follow-up)
Completed (Completed until CCO (Month 18 up to 4.5 years)) | 16 (Completed to CCO. 6 participants entered Extended Safety Follow-up, 10 participants completed Study.)
Not Completed | 9
Not completed — Transferred Back to Local Hospital | 1
Not completed — Physician and Family Decision | 1
Not completed — Transferred to Adult Services | 5
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Rituximab
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.4 (2.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 5
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 4
  Black or African American | 1
  White | 17
  Multiple | 1
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Adverse Events (AEs), Including Serious AEs
Description: An AE is any unfavourable and unintended sign (including abnormal laboratory finding), symptom, or disease temporarily associated with the use of a study drug, whether or not considered related to the study drug. A SAE is any experience that results in death, is life-threatening, requires in-patient hospitalisation or prolongation of existing hospitalisation, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is medically significant.
Time Frame: Baseline (Day 1) up to last visit (1.5-5 years)
Population: The safety population included all participants who received at least part of one infusion of rituximab.
Measure: Number; unit: percentage of participants
Groups:
- Remission Induction Phase (up to 6 Mos.) Rituximab: Participants received rituximab as an intravenous (IV) infusion of 375 milligrams per metre squared (mg/m^2) once a week on Days 1, 8, 15 and 22 during Remission Induction Phase (Day 1 (baseline) to Month 6)
- Overall Follow-up Phase (up to 4.5 Yrs) Rituximab: Participants who received rituximab during the Remission Induction Phase were followed for a minimum of 18 months during the Follow-up Phase and could receive additional rituximab or other treatments for GPA/MPA (Day 1 (baseline) up to 4.5 yrs)
Arm/Group | Remission Induction Phase (up to 6 Mos.) Rituximab | Overall Follow-up Phase (up to 4.5 Yrs) Rituximab
Number analyzed (Participants) | 25 | 25
percentage of participants
  Percentage of Participants with AEs | 100 | 100
  Percentage of Participants with SAEs | 28 | 48

2. Primary Outcome: Pharmacokinetics: Rituximab Clearance (CL)
Description: CL is a quantitative measure of the rate at which a drug substance is removed from the body. The following allometric scaling equation was used for the estimation of CL in children:
  CL= qCL X (BSA/1.9) 0.92 X 1.31*ADA
  where qCL is a typical value of clearance in millilitres per day (mL/day) for a typical participant (i.e., Body Surface Area (BSA) of 1.9 m^2 and absence of anti-rituximab antibodies (ADA)) and is equal to 258 mL/day; BSA is in m^2 and ADA is 1 when anti-rituximab antibodies are present (0 otherwise). The allometric scaling factor was 0.92. CL was calculated in millilitres per day (mL/day).
Time Frame: From Day 1 to Day 180
Population: The PK analysis population included all participants in the safety population who provided at least one evaluable PK sample.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day
Groups:
- Rituximab (Experimental): Participants received rituximab as an intravenous (IV) infusion of 375 milligrams per meter squared (mg/m^2) once a week on Days 1, 8, 15 and 22 during the Remission Induction Phase (Day 1 (baseline) to Month 6) and were followed for a minimum of 18 months (maximum 4.5yrs) during the Follow-up Phase until the Common-closeout (CCO))
Arm/Group | Rituximab (Experimental)
Number analyzed (Participants) | 25
mL/day | 204 (0.414)

3. Primary Outcome: Pharmacokinetics: Volume of Distribution (Vd) of Rituximab
Description: Vd is defined as the theoretical central volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vd was calculated in millilitres (mL).
Time Frame: From Day 1 to Day 180
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL
Arm/Group | Rituximab (Experimental)
Number analyzed (Participants) | 25
mL | 2220 (0.212)

4. Secondary Outcome: Pharmacokinetics: Area Under the Concentration-Time Curve From Time 0 to 180 Days (AUC-180) of Rituximab
Description: The AUC0-180 is a measure of the plasma concentration of rituximab over time. The AUC0-180 was calculated in micrograms per millilitres times day (mcg/mL*day).
Time Frame: From Day 1 to Day 180
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL*day
Arm/Group | Rituximab (Experimental)
Number analyzed (Participants) | 25
mcg/mL*day | 10120 (0.42)

5. Secondary Outcome: Pharmacokinetics: Maximum Plasma Concentration (Cmax) of Rituximab
Description: Cmax is the maximum observed plasma rituximab concentration. Cmax was assessed at each visit following 1st, 2nd, 3rd, and 4th IV dose of rituximab 375 mg/m^2 on Days 1, 8, 15, and 22. Cmax was calculated in micrograms per millilitre (mcg/mL).
Time Frame: From Day 1 to Day 180
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Rituximab (Experimental)
Number analyzed (Participants) | 25
mcg/mL
  1st Dose | 230 (0.166)
  2nd Dose | 305 (0.181)
  3rd Dose | 353 (0.183)
  4th Dose | 378 (0.174)

ADVERSE EVENTS:
Time Frame: Up to approximately 5 years
Description: The safety population included all participants who received at least part of one infusion of rituximab.
Groups:
- Remission Induction Phase: Rituximab: Participants received rituximab as an IV infusion of 375 mg/m^2 once a week on Days 1, 8, 15 and 22 during Remission Induction Phase (Day 1 (baseline) to Month 6)
- Overall Follow-up Phase: Rituximab: Participants who received rituximab during the remission induction phase were followed for a minimum of 18 months during the follow-up phase and could receive additional rituximab or other treatments for GPA/MPA (Day 1 (baseline) up to 4.5 yrs)
Arm/Group | Remission Induction Phase: Rituximab | Overall Follow-up Phase: Rituximab
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 7/25 | 12/25
Other Adverse Events (participants affected / at risk) | 22/25 | 24/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Remission Induction Phase: Rituximab (N=25) | Overall Follow-up Phase: Rituximab (N=25)
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 0 | 1
Sickle cell anaemia (Congenital, familial and genetic disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 1
Device related sepsis (Infections and infestations) | 0 | 1
Eye infection bacterial (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Seizure (Nervous system disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Granulomatosis with polyangiitis (Vascular disorders) | 2 | 4
Vasculitis (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Remission Induction Phase: Rituximab (N=25) | Overall Follow-up Phase: Rituximab (N=25)
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Deafness unilateral (Ear and labyrinth disorders) | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 3
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4
Constipation (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 7
Gastritis (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 4 | 5
Vomiting (Gastrointestinal disorders) | 2 | 4
Chest pain (General disorders) | 2 | 3
Non-cardiac chest pain (General disorders) | 0 | 2
Hypogammaglobulinaemia (Immune system disorders) | 0 | 3
Conjunctivitis (Infections and infestations) | 2 | 5
Ear infection (Infections and infestations) | 0 | 3
Fungal skin infection (Infections and infestations) | 0 | 2
Gastroenteritis (Infections and infestations) | 2 | 3
Herpes zoster (Infections and infestations) | 0 | 2
Influenza (Infections and infestations) | 0 | 4
Lower respiratory tract infection (Infections and infestations) | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 5
Oral herpes (Infections and infestations) | 2 | 2
Pharyngitis (Infections and infestations) | 0 | 3
Pneumonia (Infections and infestations) | 0 | 2
Sinusitis (Infections and infestations) | 0 | 3
Tooth infection (Infections and infestations) | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 4 | 12
Urinary tract infection (Infections and infestations) | 0 | 3
Viral upper respiratory tract infection (Infections and infestations) | 2 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 14 | 16
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 2
Blood immunoglobulin G decreased (Investigations) | 2 | 2
C-reactive protein increased (Investigations) | 0 | 2
Serum ferritin decreased (Investigations) | 0 | 2
Iron deficiency (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Headache (Nervous system disorders) | 4 | 9
Migraine (Nervous system disorders) | 0 | 3
Tremor (Nervous system disorders) | 2 | 2
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 0 | 2
Amenorrhoea (Reproductive system and breast disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 2
Purpura (Skin and subcutaneous tissue disorders) | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 2
Rash erythematous (Skin and subcutaneous tissue disorders) | 2 | 2
Skin striae (Skin and subcutaneous tissue disorders) | 2 | 2
Granulomatosis with polyangiitis (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 2 | 3

LIMITATIONS AND CAVEATS:
After Month 6, participants could receive treatment for GPA/MPA in accordance with local standard of care, and this could include additional rituximab infusions and/or other immunosuppressive therapies. Low participant numbers (e.g., 1 subject = 4%).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-04-26): https://cdn.clinicaltrials.gov/large-docs/97/NCT01750697/Prot_000.pdf
  • Statistical Analysis Plan (2018-09-10): https://cdn.clinicaltrials.gov/large-docs/97/NCT01750697/SAP_001.pdf